CLINICAL TRIAL: NCT01291303
Title: Optimization of Ventilator Setting by Flow and Pressure Curves Analysis During Noninvasive Ventilation for Acute Exacerbations of Chronic Obstructive Pulmonary Disease
Brief Title: Optimization of Ventilator Setting for Acute Exacerbations of Chronic Obstructive Pulmonary Disease
Acronym: NIMV01AECB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Milan (Other)
Collaborators: Ospedale Campo di Marte, UO Pneumologia e UTSIR, Lucca, IT (Unknown); Valduce Hospital (Other); IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other); Ente Ospedaliero Cantonale, Bellinzona (Other); Azienda Ospedaliera San Gerardo di Monza (Other)
Responsible Party: Dr. Fabiano Di Marco, Respiratory Unit, San Paolo Hospital, University of Milan, Milan, Italy
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NIMV01AECB
Record Dates: First submitted 2011-02-07; First posted 2011-02-08 (Estimated); Last update posted 2011-02-08 (Estimated); Status verified 2010-10

CONDITIONS: Acute Exacerbation of Chronic Obstructive Airways Disease
Keywords: Non invasive ventilation; acute exacerbation of COPD; optimized ventilation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1- optimized ventilation (Experimental): 35 COPD patients ventilated for acute exacerbations in NIV with pressure support mode.
  Interventions: Procedure: Optimized ventilation
- 2-standard setting of ventilation (Experimental): 35 COPD patients ventilated for acute exacerbations in NIV with pressure support mode.
  Interventions: Procedure: Standard ventilation

INTERVENTIONS:
Procedure: Optimized ventilation — Patients, ventilated in pressure support mode, were ventilated with initial setting PEEP and pressure support of 4 and as maximum tolerated cmH2O, inspiratory and expiratory trigger of 5 L/min and 50% of peak inspiratory flow, with changes driven by the analysis of flow and pressure curves; with a FiO2 to reach a SpO2 level between 88 and 92%.
  Arms: 1- optimized ventilation
Procedure: Standard ventilation — Patients, ventilated in pressure support mode, were ventilated with standard setting of ventilation:
  -same initial setting, same time at the bedside (15 minutes at the beginning of NIV, and 5 minutes at each patients' new evaluation) same physician that "optimized ventilation" mode, while the ventilator screen was obscured (numerical data were, however, always available).
  Arms: 2-standard setting of ventilation

SUMMARY:
The analysis of flow and pressure curves generated by ventilators can be useful in the individuation of patient-ventilator asynchrony, notably in COPD patients. To date, however, a real clinical benefit of this approach to optimize ventilator setting has not been proven. The aim of the present study was to compare: optimized ventilation, driven by the analysis of flow and pressure curves, and standard setting (same initial setting, same time at the bedside, same physician, while the ventilator screen was obscured with numerical data always available). The primary aim was the normalization of pH at two hours, whilst secondary aims were change in PaCO2, respiratory rate, patient's tolerance to ventilation (all parameter evaluated at baseline, 30, 120, 360 minutes and 24 hours after the beginning of ventilation). 70 patients (26 females, aged 78±9 years, PaCO2 74±15 mmHg, pH 7.28±0.05, mean±SD) have been enrolled, with no basal difference between the two groups.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients aged > 40 years affected by COPD exacerbation (defined as an acute change in a patient's baseline dyspnoea, cough and/or sputum beyond day-to-day variability sufficient to warrant a change in therapy), and respiratory acidosis (pH < 7.35) that were treated by NIV in addition to standard medical therapy

Exclusion Criteria:

* The needing of intubation
* The lack of informed consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-10; Primary Completion 2010-09 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
arterial pH | 2 hours
  The primary outcome was the normalization of arterial pH (=pH≥7.35) at 2 hours from the beginning of non invasive ventilation

SECONDARY OUTCOMES:
carbon dioxide tension in arterial blood (PaCO2) | 120, 360 minutes and 24 hours
  carbon dioxide tension (mmHg) in arterial blood measured 12O, 360 minutes and 24 hours after beginning of non invasive ventilation
respiratory rate (RR) | 120, 360 minutes and 24 hours after the beginning of ventilation
  respiratory rate (RR) measured 120, 360 minutes and 24 hours after the beginning of non invasive ventilation
patient's tolerance to ventilation | 30, 120, 360 minutes and 24 hours after the beginning of ventilation
  The patients tolerance to ventilation was evaluated on a visual analogue scale. This scale has been used and validated in previous studies and has five scores: 1) bad; 2) poor; 3) sufficient; 4) good; and 5) very good.
mortality | 30 days
  30-day mortality after beginning of non invasive ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Stefano Nava, MD, Study Chair — Policlinico S.Orsola Malpighi, Università di Bologna, Pneumologia e Terapia Intensiva Respiratoria Bologna, BO, Italy; Fabiano Di Marco, MD, Study Director — Respiratory Medicine Section, Dipartimento Toraco-Polmonare e Cardiocircolatorio, Università degli Studi di Milano, San Paolo Hospital
Locations (6):
- Italy (5):
  - Policlinico S.Orsola Malpighi, Università di Bologna, Pneumologia e Terapia Intensiva Respiratoria, Bologna, BO
  - Ospedale Valduce, Emergency Departement, Como, CO
  - Ospedale Campo di Marte, UO Pneumologia e UTSIR, Lucca, LU
  - Respiratory Medicine Section, Dipartimento Toraco-Polmonare e Cardiocircolatorio, Università degli Studi di Milano, San Paolo Hospital, Milan, Milan
  - Ospedale S. Gerardo, Pneumologia, Università degli Studi di Milano-Bicocca, Monza, Monza
- Ente Ospedaliero Cantonale, Intensive Care Unit, Bellinzona, Canton Ticino, Switzerland

REFERENCES:
- [Derived] Di Marco F, Centanni S, Bellone A, Messinesi G, Pesci A, Scala R, Perren A, Nava S. Optimization of ventilator setting by flow and pressure waveforms analysis during noninvasive ventilation for acute exacerbations of COPD: a multicentric randomized controlled trial. Crit Care. 2011;15(6):R283. doi: 10.1186/cc10567. Epub 2011 Nov 24. PMID 22115190